CLINICAL TRIAL: NCT03967080
Title: Adaptive Radiotherapy for High-risk Prostate Cancer Using Multiparametric MRI (ARPC-MRI) - a Feasibility Study
Brief Title: Adaptive Radiotherapy for High-risk Prostate Cancer Using Multiparametric MRI
Acronym: ARPC-MRI
Status: Completed | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RD2018-46
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This small study will investigate the feasibility of using multi-parametric MRI to introduce and support adaptive radiotherapy treatments for high-risk prostate cancer.

DETAILED DESCRIPTION:
Mount Vernon Cancer Centre at East and North Hertfordshire NHS Trust offers patients with certain cancers a treatment called adaptive radiotherapy. The aim of adaptive radiotherapy is to respond to physical changes that occur during treatment to ensure the radiation continues to be directed at the cancer and to minimise the amount of healthy tissue treated. For example, if tumour shrinkage or weight loss occurs during head and neck radiotherapy the patient may have a repeat CT scan and a new radiotherapy treatment plan after a few weeks of treatment. For patients with cancer of the bladder or cervix changes in bladder and uterus size and position can be predicted allowing the prospective creation of three radiotherapy treatment plans, each day the best fitting plan, i.e. the one that closely covers the tumour whilst giving minimal dose to normal tissues, is selected and used for treatment, this is known as plan-of-the-day adaptive radiotherapy.

Small changes in shape and position of the prostate occur but are generally the result of rectal changes which cannot be predicted, consequently adaptive radiotherapy based on physical change is not possible for prostate cancer treatments. However, recent literature suggests that magnetic resonance imaging (MRI) can detect changes within the prostate in response to radiotherapy, some studies have seen changes as early as the second week of radiotherapy treatment. A feasibility study to investigate if these changes can support radiotherapy treatment plan adaption for prostate cancer treatments is proposed, whether the plan can be adapted to give a higher treatment dose to any areas of the prostate that show poor response to radiotherapy without increasing bowel and bladder dose is of particular interest. The treatment for patients who participate in the study would not be changed but the results may help to personalise and improve the treatment of future patients.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosis of high-risk prostate cancer: any of:

   1. Gleason score of 8, 9 or 10
   2. PSA > 20
   3. T3/4
2. Patient due to receive androgen deprivation therapy (ADT)
3. Prescribed 78Gy/39# external beam radiotherapy
4. Measurable dominant intraprostatic tumour on diagnostic imaging of at least 10mm diameter
5. ≥18 years of age
6. ECOG performance status of 0-1
7. Informed, written and witnessed consent to participate is required.

Exclusion Criteria:

1. Patients who are not due to receive androgen deprivation therapy (ADT)
2. Any contraindication to MRI scanning including contraindication to MRI contrast agents
3. Previous radiotherapy to the pelvis
4. Any physical or social reasons that would make attendance for additional visits impossible.
5. Any patient with or planned for prostate fiducial markers.
6. Unable to give informed consent.
7. Patients currently enrolled in an interventional clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study looks at High-risk prostate cancer, female participants are excluded.
Study Population: 15 male patients scheduled to receive androgen deprivation therapy and external beam radiotherapy for high-risk prostate cancer at Mount Vernon Cancer Centre.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Reproducability of DW-MRI | 7 months
  Apparent diffusion coefficient (ADC)
Reproducibility of DCE-MRI | 7 months
  Using volume transfer constant
Reproducibility of DCE-MRI | 7 months
  Using leakage space as a percentage of unit volume
Reproducibility of DCE-MRI | 7 months
  Using rate constant
MP-MRI Response Correlation | 7 months
  Developing methods to identify and delineate areas of tumour according to their response to radiotherapy treatment by correlating MP-MRI kinetic parameters with anatomical T2 MRI images
Assessment of adapted dosimetry | After week 3 of radiotherapy
  Amount of acceptable radiotherapeutic dose

SECONDARY OUTCOMES:
Assessment of cell kill | 3 months
  Proportion of cells killed at given dose following androgen deprivation therapy
Tumour response prediction | 7 months
  Assess which proportion of tumours demonstrate areas of poor response that could benefit from adaptive radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Northwood, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No